CLINICAL TRIAL: NCT07062627
Title: A Pilot Study of Anbalcabtagene Autoleucel in Patients With Relapsed/Refractory Primary or Secondary Central Nervous System Lymphoma
Brief Title: Anbalcabtagene Autoleucel in Relapsed/Refractory CNS Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hyungwoo Cho (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Hyungwoo Cho, Assistant Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anbal-Cel
Record Dates: First submitted 2025-05-27; First posted 2025-07-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Primary CNS Lymphoma (PCNSL); Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: lymphoma; CAR-T; Anbalcabtagene autoleucel
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anbal-Cel arm (Experimental): Anbal-cel will be administered as a single intravenous infusion on Day 1, within 30 minutes of thawing.
  The intended dose is 2 × 10⁶ CAR-T cells/kg, with a maximum of 2 × 10⁸ cells.
  Interventions: Genetic: Anbal-cel

INTERVENTIONS:
Genetic: Anbal-cel — On Day 1 (D1), Anbal-cel will be administered only to subjects who meet the final inclusion/exclusion criteria for Anbal-cel administration before the infusion.
  As premedication before Anbal-cel administration, acetaminophen or paracetamol, and diphenhydramine or H1 antihistamine will be given.
  Anbal-cel will be administered as a single intravenous infusion on Day 1 within 30 minutes of thawing, at the dose presented in the following table:
  Dose: 2x10^6 (CAR-T cells/kg)* Maximum 2 x 10^8 cells

SUMMARY:
This clinical study aims to evaluate the tolerability, safety, and efficacy of Anbal-cel in patients with recurrent or refractory PCNSL or SCNSL.

Subjects who have provided written consent and meet the inclusion and exclusion criteria through screening evaluations will undergo leukapheresis (LP) for Anbal-cel manufacturing. Subjects whose collected nucleated cells are confirmed suitable for Anbal-cel production will be enrolled in the clinical study.

Prior to Anbal-cel administration, lymphodepletion therapy will be performed and must be completed at least 2 days before Anbal-cel administration. Anbal-cel will be administered to subjects who meet the inclusion and exclusion criteria for Anbal-cel administration.

Study subjects will be hospitalized for a minimum of 7 days to closely monitor adverse events and receive prompt necessary treatment after Anbal-cel administration. All study subjects will undergo primary visit evaluations for 12 months following Anbal-cel administration.

Subjects who discontinue primary visit evaluations before the 12-month visit will undergo an end of study 1 (EOS1) visit for safety observation. For subjects whose primary visit evaluations end before the 12-month visit due to disease progression (PD), withdrawal of consent for primary visit evaluations, or subsequent anti-cancer therapy, secondary follow-up visits will be conducted from the EOS1 visit to the 12-month time point (EOS2). The timing of the first secondary follow-up visit will be determined based on when the subject's primary visit evaluation was discontinued.

A separate long-term follow-up study is planned to monitor long-term safety, including delayed adverse events (AEs), in subjects who received Anbal-cel. In this long-term follow-up study, each subject will be followed for 15 years from the date of Anbal-cel administration. All specific details, including the visit schedule and examination items for the long-term follow-up study, will be described in a separate protocol.

DETAILED DESCRIPTION:
Primary central nervous system lymphoma (PCNSL) and secondary CNS lymphoma (SCNSL) are rare and aggressive subtypes of non-Hodgkin lymphoma (NHL) with poor prognoses in relapsed or refractory cases. Existing salvage therapies provide limited clinical benefit due to low response durability and high relapse rates, underscoring the need for novel therapeutic strategies.

Chimeric antigen receptor T (CAR-T) cell therapy is a form of adoptive cell transfer (ACT) that reprograms T cells to target specific tumor antigens via genetically engineered immunoreceptors. Unlike T-cell receptor (TCR)-based approaches, CAR-T cells recognize tumor-associated antigens independently of HLA presentation.

Anbalcabtagene autoleucel (Anbal-cel) is an investigational autologous anti-CD19 CAR-T cell product, incorporating a CD19-specific scFv, CD8 hinge and transmembrane domains, a 4-1BB co-stimulatory domain, and a CD3-zeta signaling domain. Upon CD19 engagement, Anbal-cel forms an immunological synapse and triggers effector functions, including proliferation, cytokine secretion (e.g., IFN-γ, IL-6, TNF-α, GM-CSF), and cytotoxic activity via perforin/granzyme and death receptor pathways.

Notably, Anbal-cel is engineered to minimize T-cell exhaustion by downregulating immune checkpoint molecules such as PD-1 and TIGIT, which are frequently overexpressed in B-cell lymphoma. This design is anticipated to enhance antitumor efficacy relative to conventional anti-CD19 CAR-T therapies.

This single-arm, open-label pilot study aims to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of Anbal-cel in patients with relapsed or refractory PCNSL and SCNSL. In the prior phase 1/2 study (CRC01-01, NCT04836507), patients with CNS involvement were excluded; this study represents the first clinical evaluation of Anbal-cel in this population.

The study includes a safety lead-in phase involving an initial cohort of three patients receiving the recommended phase 2 dose (RP2D) of 2 × 10⁶ CAR-T cells/kg. A Safety Review Committee (SRC) will assess initial safety data before proceeding with additional enrollment.

To prepare for Anbal-cel infusion, patients will receive a lymphodepletion regimen of fludarabine (30 mg/m²/day) and cyclophosphamide (500 mg/m²/day) on Days -5 to -2. This approach is supported by prior CAR-T studies (e.g., Yescarta®), which demonstrated improved expansion and persistence with acceptable safety profiles.

The **primary objective** is to assess the overall response rate (ORR) using the International Primary CNS Lymphoma Collaborative Group criteria.

* Secondary objectives** include:

  * Complete response rate (CRR)
  * Time to response (TTR)
  * Duration of response (DOR)
  * Event-free survival (EFS)
  * Progression-free survival (PFS)
  * Overall survival (OS)
  * Safety and tolerability
  * Pharmacokinetics and immune profiling
* Exploratory objectives** include evaluating associations between Anbal-cel expansion, cytokine levels, and immune-related adverse events (e.g., CRS, ICANS), as well as biomarker analyses (e.g., CD19, PD-1, TIGIT, LAG-3, TIM-3 in tumor or CSF) to characterize immune phenotype and gene expression changes linked to response.

All patients will undergo long-term follow-up for 5 years in accordance with gene therapy guidance. Additionally, subjects who provide consent will be enrolled in a separate 15-year long-term safety follow-up protocol. Dose adjustments and WBC thresholds will guide lymphodepletion decisions based on patient condition and clinical safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 years or older who voluntarily agree to participate in this clinical study and provide written consent.
2. Patients with recurrent/refractory B-cell lymphoma confirmed histologically according to the 2017 WHO classification, and who meet one of the following conditions:

   Primary central nervous system lymphoma (PCNSL) of the DLBCL subtype Secondary central nervous system involvement of DLBCL with no involvement outside the central nervous system
3. Patients who failed treatment with a previous regimen that included high-dose methotrexate or patients intolerant to high-dose methotrexate.
4. Patients who agree to provide tumor tissue. If a stored tumor tissue sample is available, it can be submitted only if it was collected within 6 months prior to participation in the clinical study and if no systemic anticancer treatment was administered after collection. If the stored tissue sample does not meet these conditions, tumor tissue must be obtained through a core needle biopsy or excisional biopsy during the screening period. If the investigator deems the biopsy to be medically unsafe for the patient, the decision on whether to enroll the patient in the clinical study can be made in consultation with the patient's clinical physician.
5. Individuals with an ECOG performance status score of 2 or lower at the time of screening.
6. Individuals with appropriate renal and liver function confirmed by laboratory test results:

   Total Bilirubin ≤2.0 mg/dL (for individuals with Gilbert-Meulengracht syndrome: total bilirubin ≤3.0 × upper limit of normal (ULN), direct bilirubin ≤1.5 x ULN) Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 × ULN (if liver metastasis is confirmed: AST, ALT ≤5 × ULN) Serum creatinine ≤1.5 x ULN Estimated glomerular filtration rate (eGFR)* ≥60 mL/min/1.73 m²

   *MDRD-GFR (mL/min/1.73 m²) = 186 × (serum creatinine)-1.154 × (age)-0.203 (× 0.742 for females)
7. Individuals with appropriate hematologic function confirmed within 2 weeks prior to screening without transfusion, based on the following criteria:

   Hemoglobin >8.0 g/dL Absolute neutrophil count (ANC) >1,000/μL Absolute lymphocyte count (ALC) ≥300/μL Platelets ≥50,000/μL
8. Individuals who are hemodynamically stable at the time of screening, have no signs of pericardial effusion, and have a left ventricular ejection fraction of 50% or higher based on an echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
9. Individuals from whom adequate non-mobilized cells for Anbal-cel manufacturing can be collected through leukapheresis.
10. Individuals with an expected survival of 12 weeks or longer.
11. Individuals who agree to comply with the scheduled site visits, examination schedules, and assessments as per the protocol during the course of the clinical study, including primary and secondary follow-up visits.
12. Women of childbearing potential and men who agree to use appropriate contraception* for at least 12 months after Anbal-cel administration until Anbal-cel is no longer detected in PCR tests. *Hormonal contraception, intrauterine system implants, dual barrier methods (simultaneous use of a diaphragm or cervical cap with a condom and spermicide), sterilization procedures (e.g., vasectomy, bilateral tubal ligation), etc.

Exclusion Criteria:

1. Individuals with a history of allogeneic hematopoietic stem cell transplantation.
2. Individuals with the following medical history:

   * History of other malignancies, except B-cell non-Hodgkin lymphoma, within 3 years prior to screening (however, individuals with a history of basal cell carcinoma, squamous cell carcinoma of the skin, localized prostate cancer, papillary thyroid cancer, cervical carcinoma in situ, or early-stage gastric cancer may participate if the investigator considers them to be fully cured after successful treatment, even if 3 years have not passed).
   * History of unstable angina and/or myocardial infarction within 12 months prior to screening.
   * History of thromboembolism, pulmonary embolism, or bleeding diatheses within 6 months prior to screening.
   * History of hypoxia, clinically significant pleural effusion, or abnormal electrocardiogram findings within 6 months prior to screening.
3. Individuals with the following conditions at the time of screening:

   * Known positive for human immunodeficiency virus (HIV).
   * Active neurological autoimmune or inflammatory diseases (e.g., Guillain-Barré syndrome, amyotrophic lateral sclerosis).
   * Recurrent or symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response despite treatment in the 3 months prior to screening.
4. Individuals whose disease is rapidly progressing, as determined by the investigator.
5. Individuals who have undergone major surgery requiring general anesthesia or respiratory support within 4 weeks prior to screening (however, video-assisted thoracoscopic surgery (VATS) or open-and-closed (ONC) surgery is permissible if conducted within 2 weeks).
6. Individuals with severe infections requiring the administration of antibiotics, antifungals, or antivirals at the time of screening or with uncontrolled active infections.
7. Individuals who have received or been exposed to other investigational drugs or devices within 4 weeks prior to screening.
8. Pregnant or breastfeeding women.
9. Individuals with a hypersensitivity to the ingredients of the investigational drug.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) of Anbal-cel, as determined according to the International Primary CNS Lymphoma Collaborative Group. | 24 months
  The objective response rate (ORR) is defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR), as assessed by the investigator. Subjects who do not achieve CR or PR will be considered non-responders in the analysis.

SECONDARY OUTCOMES:
Complete response rate (CRR) | 24 months
  The Complete Response Rate (CRR) is defined as the proportion of patients who achieve a complete response (CR) as their best overall response during the study period. CR is determined according to the International Primary CNS Lymphoma Collaborative Group.
time to response, TTR | 24 months
  Defined as the time from the date of Anbal-cel administration to the date when complete response (CR) or partial response (PR) is first documented.
Duration of response (DOR) | 24 months
  This analysis will be conducted in subjects who achieve complete response (CR) or partial response (PR). Duration is defined as the time from the first documentation of CR or PR to the earliest occurrence of disease progression (PD), relapse, or death due to the study disease. Survival probability and 95% confidence intervals will be estimated using the Kaplan-Meier method.
Event-free survival (EFS) | 24 months
  Defined as the time from the date of Anbal-cel administration to the earliest occurrence of disease progression (PD), relapse, initiation of subsequent anti-cancer therapy, or death. The median survival time and two-sided 95% confidence intervals will be estimated by treatment group using the Kaplan-Meier method.
Progression-free survival (PFS) | 24 months
  Defined as the time from the date of Anbal-cel administration to the earliest occurrence of disease progression (PD), relapse, or death. The median survival time and two-sided 95% confidence intervals will be estimated by treatment group using the Kaplan-Meier method.
Overall survival (OS) | 24 months
  Defined as the time from the date of Anbal-cel administration to death from any cause. The median survival time and two-sided 95% confidence intervals will be estimated by treatment group using the Kaplan-Meier method.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During 24 months
  Severity of adverse events will be graded by NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events) v5.0
Evaluation of the pharmacokinetic properties of Anbal-cel | 24 months
  PK parameters include Maximum Plasma Concentration (Cmax, Peak Plasma Concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Hyungwoo Cho, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No